CLINICAL TRIAL: NCT07332208
Title: Evaluation of Breastfeeding Education Delivered Using the Role-Play Technique Among Adolescent Pregnant Women: A Randomized Controlled Study
Brief Title: Evaluation of Breastfeeding Education Using the Role-Play Technique
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Ayşegül Ciftçiler, Graduate Researcher, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025/019 Ethics Committee Appr
Record Dates: First submitted 2025-12-24; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Nursing Education; Breastfeeding Education; Adolescent Pregnancy; Nursing Interventions
Keywords: Breastfeeding; Adolescent Pregnancy; Breastfeeding Education; Role-play education
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either an intervention group receiving role-play-based breastfeeding education or a control group receiving routine care. Outcomes are compared between parallel groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adolescent Pregnant Women Receiving Standard Breastfeeding Education (Active Comparator): Participants in this cohort receive standard breastfeeding education as part of routine prenatal care. The education is delivered using conventional instructional methods and does not include the role-play technique.
  Interventions: Other: Standard Breastfeeding Education
- Adolescent Pregnant Women Receiving Role-Play-Based Breastfeeding Education (Experimental): Participants in this cohort receive breastfeeding education delivered using the role-play technique as part of prenatal care. The intervention includes interactive role-play scenarios designed to improve breastfeeding knowledge, skills, and self-efficacy.
  Interventions: Behavioral: Role-Play-Based Breastfeeding Education

INTERVENTIONS:
Other: Standard Breastfeeding Education — Participants receive standard breastfeeding education delivered according to routine prenatal care practices using conventional instructional methods.
  Arms: Adolescent Pregnant Women Receiving Standard Breastfeeding Education
Behavioral: Role-Play-Based Breastfeeding Education — Participants receive breastfeeding education delivered using role-play techniques as part of routine prenatal care. The intervention includes interactive role-play scenarios designed to improve breastfeeding knowledge, practical skills, and breastfeeding self-efficacy.
  Arms: Adolescent Pregnant Women Receiving Role-Play-Based Breastfeeding Education

SUMMARY:
Adolescence is defined as a period of rapid biological and physical development, as well as sexual and psychosocial maturation, during which the individual gains independence and social productivity. This developmental period largely corresponds to the age range of 10 to 19 years, consistent with the WHO (World Health Organization) definition of adolescence. Adolescent pregnancy is considered a public health issue by the WHO due to its biopsychosocial effects on maternal and child health. Adolescents often seek antenatal care late due to a lack of information, limited access to healthcare, social pressure, and fear of stigma. There are many increased risks for both mother and newborn during adolescent pregnancy. The low educational level of adolescent pregnant women also negatively affects access to necessary healthcare services. Breastfeeding is the most appropriate way to provide breast milk to the baby for healthy development. It is the healthiest, easiest, most natural, and most economical method of feeding the baby. The World Health Organization (WHO) recommends initiating breastfeeding within the first hour after birth . Providing planned education to protect and improve the health of individuals, families, and communities, and to ensure they acquire correct health behaviors, is among the fundamental duties of nurses, who are in the most contact with healthy/sick individuals in the community.

Role-playing is among the educational methods used to increase awareness in nursing. Role-playing is used in education as a skill-oriented teaching method that enables social communication skills, active listening, empathy for emotions, and seeing excerpts from real life in teaching knowledge and skills. Especially in educational groups with low education levels, the effectiveness of education can be increased by using the role-playing technique.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent pregnant women
* Not having received any formal breastfeeding education previously

Exclusion Criteria:

* Pregnant women outside the adolescent age range
* Having previously received breastfeeding education

Ages: 16 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Knowledge Level | Baseline (pre-intervention) and immediately after the intervention
  Change in breastfeeding knowledge level assessed using a structured questionnaire developed to evaluate breastfeeding-related knowledge.

SECONDARY OUTCOMES:
Breastfeeding Self-Efficacy Level | Baseline (pre-intervention) and immediately after the intervention
  Change in breastfeeding self-efficacy level assessed using the Prenatal Breastfeeding Self-Efficacy Scale (PBSES). The scale evaluates mothers' confidence in their ability to breastfeed.

CONTACTS AND LOCATIONS:
Locations (1):
- Şanlıurfa Eyyübiye Ilçe Sağlık Müdürlüğü, Sanliurfa, Şanlıurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and institutional restrictions and to protect participant confidentiality.